CLINICAL TRIAL: NCT01776801
Title: Assessment of Autonomic Neuronal Changes During Moderate Rise of Intracranial Pressure in Human
Acronym: CESNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 07 299 03
Record Dates: First submitted 2013-01-23; First posted 2013-01-28 (Estimated); Last update posted 2013-02-25 (Estimated); Status verified 2013-02

CONDITIONS: Increased Intracranial Pressure Disorders
Keywords: intracranial baroreflex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydrocephalus (Experimental): Patients suffering of hydrocephalus (cognitive impairment, gait disturbance, urinary incontinence and enlargement of the ventricles) require for clinical purpose infusion studies i.e. injection of mock cerebrospinal fluid (CSF) in the sub arachnoid space to artificially increase ICP. We aim at using infusion studies as a indirect tool to assess whether a moderate increase in ICP has any influence on haemodynamics.
  Interventions: Other: Infusion

INTERVENTIONS:
Other: Infusion — Infusion studies are performed in daily clinical routine to measure cerebrospinal fluid resistance outflow. During this test ICP is slowly and securely raised. Investigators plan to analyze what are the consequences of this ICP rise in terms of autonomic system and hemodynamics.

SUMMARY:
The purpose of this project is to determine during moderate rise of intracranial pressure (ICP) in awake patient, the change in autonomic function and its influence on cerebral and systemic haemodynamics.

DETAILED DESCRIPTION:
From preliminary data, we know that changes in ICP influences both systemic and cerebral haemodynamics, introducing the concept of intracranial baroreflex We have to i) confirm the presence of this intracranial baroreflex, ii) analyze the changes in autonomic function during moderate rise in intracranial pressure (ICP) in human, and iii) correlate the changes in cerebral and systemic haemodynamics with autonomic function.

ELIGIBILITY:
Inclusion Criteria:

* patient suspect of hydrocephalus with gait problems, urine incontinence and mild cognitive impairment.
* signed consent

Exclusion Criteria:

* psychiatric problems
* severe cognitive decline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-01; Primary Completion 2011-05 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
change in sympathetic nerve activity after rise in ICP | within few minutes
  Assessment of autonomic neural function using.
  1. microneurography to assess the muscle sympathetic nerve activity
  2. measurement of the plasma level changes of noradrenaline
  3. power spectral analysis of heart rate and arterial blood pressure

SECONDARY OUTCOMES:
change in hemodynamics after rise in ICP | within few minutes
  Assessment of haemodynamics
  1. Cerebral haemodynamics. using Transcranial doppler
  2. Systemic haemodynamics measured with photoplethysmography

CONTACTS AND LOCATIONS:
Overall Officials: Eric SCHMIDT, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (3):
- France (3):
  - University Hospital of Toulouse, Toulouse, France
  - University Hospital Toulouse, Toulouse
  - University Hospital, Toulouse